CLINICAL TRIAL: NCT02678793
Title: An Open-Label, Multiple-Dose Extension Study to Evaluate the Safety and Efficacy of CNTX-4975 in Subjects With Painful Intermetatarsal Neuroma (Morton's Neuroma)
Brief Title: A Study to Evaluate the Safety and Efficacy of CNTX-4975 in Subjects With Painful Intermetatarsal Neuroma (Morton's Neuroma)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centrexion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4975-MN-203
Record Dates: First submitted 2016-01-18; First posted 2016-02-10 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Morton's Neuroma
MeSH Terms: conditions — Morton Neuroma | interventions — CNTX-4975

ARMS (1):
- Subjects who have completed Study 4975-MN-202 will be eligible (Other): Subjects who have completed Study 4975-MN-202 will be eligible to receive open-label treatment with CNTX-4975 200 μg in Study 4975-MN-203 if they meet the inclusion/exclusion criteria.
  Interventions: Drug: CNTX-4975

INTERVENTIONS:
Drug: CNTX-4975

SUMMARY:
Subjects who have completed study 4975-MN-202 will be eligible to receive open-label treatment with CNTX-4975 200 µg in study 4975-MN-203 if they meet the inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged >18 years at the time of the Screening Visit.
2. Completion of study 4975-MN-202.
3. Female not of childbearing potential, defined as post-menopausal for at least 1 year, or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or practicing one of the following medically acceptable methods of birth control throughout the study period:

   1. Hormonal methods such as oral, implantable, injectable, or transdermal contraceptives for a minimum of 1 full cycle (based on the subject's usual menstrual cycle period) before investigational product (IP) administration.
   2. Total abstinence from sexual intercourse since the last menses before IP administration.
   3. Intrauterine device.
   4. Double barrier method (condoms, sponge, diaphragm, with spermicidal jellies or cream).
4. Willing and able to understand the study requirements, abide by the study restrictions, complete the study procedures, pain scales, and weekly IWRS/IVRS entries, and to communicate meaningfully with the study personnel.
5. Signed an Informed Consent Form approved by the Institutional Review Board.
6. Subject agrees to take only the rescue medications for neuroma foot pain from the time of screening through study completion, and agrees to discontinue all topical medications for neuroma pain after Screening.

Exclusion Criteria:

1. Other chronic pain anywhere in the body that is severe in intensity or would interfere with the subject's ability to evaluate foot pain from intermetatarsal neuroma.
2. Signs of arterial insufficiency in the feet, including clinically meaningful edema.
3. Raynaud's disease or phenomenon, previous frostbite, or other cause of vascular instability in the feet resulting from application of cold to the foot.
4. Daily use of opioids for any condition.
5. Corticosteroid injection in the affected foot within 30 days of Screening.
6. Presence of any medical condition (or taking any medication) or unstable health status that, in the judgment of the investigator, might adversely impact the conduct of the study or resulting data, including chronic conditions that are likely to alter the rate of healing or are likely to result in safety complications unrelated to the study medication, such as uncontrolled diabetes mellitus or vascular disease.
7. Clinically significant abnormal laboratory result at the Screening Visit (in the opinion of the investigator).
8. Has a positive pregnancy test at the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of repeat injections of CNTX-4975 through assessment of incidence, intensity, relationship and seriousness of treatment-emergent adverse events | over the course of 1 year.
Evaluate the safety and tolerability of repeat injections of CNTX-4975 through treatment-emergent changes in vital signs and laboratory tests | over the course of 1 year.

SECONDARY OUTCOMES:
To evaluate the analgesic efficacy of repeat doses of CNTX-4975 by change in NPRS. | over the course of 1 year.
To evaluate the analgesic efficacy of repeat doses of CNTX-4975 by change in Patient Global Impression of Change | over the course of 1 year.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Arizona Research Center, Phoenix, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - TriWest Research Associates, LLC, El Cajon, California
  - Chesapeake Research Group, Pasadena, Maryland
  - Center for Advanced Medicine & Research, City of Saint Peters, Missouri
  - University Orthopedics Center, Altoona, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Allcare Foot and Ankle Centre, Arlington, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - The Education & Research Foundation, Inc., Lynchburg, Virginia